CLINICAL TRIAL: NCT02310542
Title: Comparison of Two Extracorporeal Liver Support System (With or Without Recirculation) : MARS (Molecular Adsorbents Recirculating System) Versus SPAD (Single Pass Albumin Dialysis) in Severe Liver Failure.
Brief Title: Comparison of Two Liver Dialysis Systems : MARS Versus SPAD in Severe Liver Failure
Acronym: MARSPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010.652
Record Dates: First submitted 2014-11-14; First posted 2014-12-08 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Liver Failure, Acute; Chronic Hepatic Failure
MeSH Terms: conditions — Liver Failure, Acute; End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MARS-SPAD (Experimental): Patients will receive first the MARS albumin dialysis system and then, in a second time, the SPAD albumin dialysis system.
  Interventions: Device: MARS albumin dialysis system; Device: SPAD albumin dialysis system
- SPAD-MARS (Experimental): Patients will receive first the SPAD albumin dialysis system and then, in a second time, the MARS albumin dialysis system.
  Interventions: Device: MARS albumin dialysis system; Device: SPAD albumin dialysis system

INTERVENTIONS:
Device: MARS albumin dialysis system
Device: SPAD albumin dialysis system

SUMMARY:
A critical issue of the clinical syndrome in liver failure is the accumulation of toxins not cleared by the failing liver. Based on this hypothesis, albumin dialysis is used to remove those substances. Albumin dialysis with recirculation (MARS) is the most used system but required specific system and expert environment. Alternative system without recirculation (SPAD) is less expensive and can be realised in critical care services trained to extrarenal epuration. The primary objective of this study is to compare biological and clinical efficacy, pulsatility index of middle cerebral artery modification and tolerance of both systems.

This is a prospective, open, cross-over comparative study of two albumin dialysis system. Each patient will receive the two systems in an randomly assessed order. Patients are divided up according to bilirubin plasmatic level. (250µmol/L to 400 µmol/L and >400µmol/L).

ELIGIBILITY:
Inclusion Criteria:

* severe hepatic failure on acute liver failure or acute on chronic liver failure
* hyperbilirubinemia (total plasmatic bilirubin level above 250µmol/L)
* hepatic encephalopathy or pruritus or hepatorenal syndrome.
* waiting for liver function recovery or liver transplantation
* Signed written informed consent by patient or patient's legally appointed representative or reliable person
* affiliation to social security

Exclusion Criteria:

* contraindication to extra-renal epuration
* hypersensibility to albumin or excipients
* patients for whom 2 albumin dialysis treatment cannot be considered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-12; Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Comparison of total plasmatic bilirubin level before and after two albumin dialysis systems : with recirculation (MARS™ system) and without recirculation (SPAD™ system) | Before and at the end of a MARS™ dialysis (8h) and before and at the end of a SPAD™ system dialysis (10h). Participants will be followed for the duration of critical care stay, an expected average of 1 week
  Determination of total plasmatic bilirubin level will be performed by arterial sample and expressed in µmol/liter. Total plasmatic bilirubin purification will be compared between the two dialysis systems: total plasmatic bilirubin level will be measured before and at the end of MARS™ dialysis (8 hours) and before and at the end of SPAD™ dialysis (10 hours) ; the two variations will be compared. Each patient will receive the two dialysis systems separated by a free interval that will last between 12 and 48 hours.

SECONDARY OUTCOMES:
Comparison of bile acids and conjugated bilirubin levels before and after two albumin dialysis systems: with recirculation (MARS™ system) and without recirculation (SPAD™ system). | Before and at the end of a MARS™ system dialysis (8h) and before and at the end of a SPAD™ dialysis (10h) . Participants will be followed for the duration of critical care stay, an expected average of 1 week.
  Determination of bile acids and conjugated bilirubin levels will be performed by arterial sample and expressed in µmol/liter. Bile acids and conjugated bilirubin purifications will be compared between the two dialysis systems: Bile acids and conjugated bilirubin levels will be measured before and at the end of MARS™ dialysis (8 hours) and before and at the end of SPAD™ dialysis (10 hours) ; the two variations will be compared. Each patient will receive the two dialysis systems separated by a free interval that will last between 12 and 48 hours.
Comparison of hepatic encephalopathy score before and after two albumin dialysis systems : with recirculation (MARS™ system) and without recirculation (SPAD™ system) | Before and at the end of a MARS™ system dialysis (8h) and before and at the end of a SPAD™ system dialysis (10h) . Participants will be followed for the duration of critical care stay, an expected average of 1 week.
  Determination of hepatic encephalopathy score will be performed by clinical evaluation. Hepatic encephalopathy score will be compared between the two dialysis systems: hepatic encephalopathy score will be measured before and at the end of MARS™ dialysis (8 hours) and before and at the end of SPAD™ dialysis (10 hours) ; the two variations will be compared. Each patient will receive the two dialysis systems separated by a free interval that will last between 12 and 48 hours.
Comparison of pulsatility index of middle cerebral artery recorded by transcranial doppler before and after two albumin dialysis system : with recirculation (MARS™ system) and without recirculation (SPAD™ system) | Before and at the end of a MARS™ dialysis (8h) and before and at the end of a SPAD™ system dialysis (10h). Participants will be followed for the duration of critical care stay, an expected average of 1 week
  Pulsatility index of middle cerebral artery will be recorded by transcranial doppler. Pulsatility index of middle cerebral artery will be compared between the two dialysis systems: Pulsatility index of middle cerebral artery will be measured before and at the end of MARS™ dialysis (8 hours) and before and at the end of SPAD™ dialysis (10 hours) ; the two variations will be compared. Each patient will receive the two dialysis systems separated by a free interval that will last between 12 and 48 hours.
Comparison of tolerance of two albumin dialysis sytems : with recirculation (MARS™ system) and without recirculation (SPAD™ system) | During MARS™ system dialysis (8h) and during SPAD™ system dialysis (10h) . Participants will be followed for the duration of critical care stay, an expected average of 1 week.
  Tolerance will be evaluated by effect of albumin dialysis on coagulation indices : prothrombin time (seconds) and international normalized ratio, activated partial thromboplastin time ratio, fibrinogen level (g/L), factor V level (%), platelet count (×10(9) /L), hemoglobin level (g/L), red cell count (10(12)/L), hematocrit level (%). Coagulation indices will be measured by an arterial sample before and at the end of MARS™ dialysis (8 hours) and before and at the end of SPAD™ dialysis (10 hours) ; the two variations will be compared. Each patient will receive the two dialysis systems separated by a free interval that will last between 12 and 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Serge Duperret, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix Rousse - Service de réanimation chirurgicale, Lyon, France

REFERENCES:
- [Result] Wallon G, Guth C, Guichon C, Thevenon S, Gazon M, Viale JP, Schoeffler M, Duperret S, Aubrun F. Extracorporeal Albumin Dialysis in Liver Failure with MARS and SPAD: A Randomized Crossover Trial. Blood Purif. 2022;51(3):243-250. doi: 10.1159/000515825. Epub 2021 Jun 17. PMID 34139706